CLINICAL TRIAL: NCT05066256
Title: Left Ventricular Diastolic Function Compare to Inferior Vena Cava Diameter Variation as Predictor of Fluid Responsiveness in Mechanical Ventilated Patients With Shock
Brief Title: LV Diastolic Function vs IVC Diameter Variation as Predictor of Fluid Responsiveness in Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Si 752/2020
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Shock; Septic Shock
Keywords: shock; fluid responsiveness; left ventricular diastolic dysfunction; Mitral E/e'
MeSH Terms: conditions — Shock; Shock, Septic; Ventricular Dysfunction, Left

STUDY DESIGN:
Intervention Model Description: Pre-experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluid responsive test (Experimental): Measure cardiac output, inferior vena cava (IVC) diameter variation and LV diastolic function (E/e') baseline Fluid challenge Measure cardiac output, IVC diameter variation and LV diastolic function (E/e') after fluid challenge
  Interventions: Diagnostic Test: Left ventricular diastolic function; Diagnostic Test: Inferior vena cava variation

INTERVENTIONS:
Diagnostic Test: Left ventricular diastolic function — Transthoracic echocardiography Mitral E/e'
  Other Names: Mitral E/e'
Diagnostic Test: Inferior vena cava variation — Inferior vena cava variation from ultrasound
  Other Names: IVC variation

SUMMARY:
Fluid responsive is defined as increasing in Cardiac output or Stroke volume by 10-15% after fluid challenge. Left ventricular diastolic dysfunction is associated with lower left ventricular end-diastolic volume (LVEDV) resulting in a less cardiac output increment after fluid challenge. However, Left ventricular diastolic function indicated by the Mitral E/e' ratio from transthoracic echocardiography, was rarely studied for fluid responsiveness evaluation.

DETAILED DESCRIPTION:
Fluid therapy is one of the main treatments in patients with shock to increase Oxygen delivery by increasing Cardiac output or Stroke volume. However excess fluid intake may cause fluid overload, resulting in tissue edema, lung edema and organ dysfunction, which can lead to patient deterioration.

Fluid responsiveness, defined as increasing in Cardiac output or Stroke volume by 10-15% after fluid challenge, is being recommended to evaluate in-patients with shock, according to European Society of Intensive Care Medicine (ESICM). Cardiac output measurement is often invasive or requires an expensive device, therefore, tests for predicting fluid responsiveness have been used to substitute direct Cardiac output measurement.

Left ventricular diastolic dysfunction is associated with a decreasing Left ventricular end-diastolic volume, resulting in a less cardiac output increment after fluid challenge and can be measured by using Mitral E/e' ratio via transthoracic echocardiography.

Despite being a non-invasive test, the Mitral E/e' ratio obtained from Echocardiography was rarely studied for the prediction of fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* Diagnosis of shock defined by systolic blood pressure < 90 mmHg or mean arterial blood pressure < 65 mmHg and/or clinical hypoperfusion
* Mechanically ventilated without ventilator dyssynchrony and no ventilator triggering
* Present of central venous cather or arterial catheter

Exclusion Criteria:

* Age < 18 years
* Frankly hypovolemic shock or hemorrhagic shock
* Suspicious of cardiogenic shock
* Suspicious of acute decompensated heart failure
* Suspicious of acute coronary syndrome
* Denied participation or denied inform consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Fluid responsiveness | 6 hours
  Fluid responsiveness defined by increase in cardiac output at least 15% or increase in systolic blood pressure at least 10 mmHg or increase in mean arterial pressure at least 5 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Surat Tongyoo, Principal Investigator — Mahidol University
Locations (1):
- Department of Medicine, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Anonymus participant data will be available after request with ethical committee approval.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within 6 months after study publication
Access Criteria: Request to principal investigator after ethical committee approval